CLINICAL TRIAL: NCT00003140
Title: A Phase III Randomized Double Blind Study of Letrozole Versus Placebo in Women With Primary Breast Cancer Completing Five or More Years of Adjuvant Tamoxifen
Brief Title: Letrozole After Tamoxifen in Treating Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); North Central Cancer Treatment Group (Network); ETOP IBCSG Partners Foundation (Network); Eastern Cooperative Oncology Group (Network); SWOG Cancer Research Network (Network); Cancer and Leukemia Group B (Network); European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MA17; U10CA025224 (NIH); CAN-NCIC-MA17 (Registry Identifier: PDQ); CALGB-49805; E-JMA17; EORTC-10983; IBCSG-BIG97-01; NCCTG-JMA17; SWOG-JMA17; JRF-Vor-Int-10; NCCTG-CAN-MA17; SWOG-CAN-MA17; CDR0000065921 (Other: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral letrozole once daily.
  Interventions: Drug: letrozole
- Arm II (Placebo Comparator): Patients receive oral placebo once daily.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: letrozole — Given orally
  Other Names: Femara
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using letrozole may fight breast cancer by reducing the production of estrogen.

PURPOSE: This randomized phase III trial is studying letrozole to see how well it works in treating women with breast cancer who have received tamoxifen for at least 5 years.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the disease-free survival and overall survival of postmenopausal women with primary breast cancer who have completed at least five years of adjuvant aromatase inhibitor as initial therapy or after tamoxifen treated with letrozole or placebo.

Secondary

* Compare the incidence of contralateral breast cancer in patients treated with these regimens.
* Evaluate the long-term clinical and laboratory safety of letrozole, in terms of lipid profile, cardiovascular morbidity and mortality, incidence of bone fractures, change in bone density, and common toxic effects, in this patient population.
* Compare the quality of life of patients treated with these regimens. Re-randomization

Primary

* Compare disease-free survival of patients who, after receiving at least 4.5 years of letrozole, are re-randomized to receive an additional 5 years of letrozole vs placebo.

Secondary

* Determine whether common genetic polymorphisms for genes encoding proteins involved in pharmacokinetic and/or pharmacodynamic pathways for letrozole contribute to individual variation in toxicity and efficacy of letrozole therapy.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to receptor status (positive vs unknown), lymph node status (negative vs positive vs unknown), prior adjuvant chemotherapy (yes vs no), interval between last dose of aromatase inhibitor therapy and randomization (< 6 months vs 6 months-2 years), and duration of prior tamoxifen use (0 years vs < 2 years vs 2-4.5 years vs > 4.5 years). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral letrozole once daily.
* Arm II: Patients receive oral placebo once daily. In both arms, treatment continues for 5 years in the absence of disease progression or unacceptable toxicity. Patients in arm II may then be offered oral letrozole once daily for up to 5 years.

Quality of life is assessed at baseline, at 6 months, and then annually for 4.5 years.

* Double-blind, re-randomization:

Patients who complete ≥ 4.5 years of letrozole (arm I) and who did not experience recurrent disease or new primary breast cancer, including ductal carcinoma in situ, may participate in the double-blind, placebo-controlled, re-randomization portion of the study. Patients are stratified according to lymph node status at enrollment (negative vs positive vs unknown), prior adjuvant chemotherapy (yes vs no), and interval between last dose of letrozole and re-randomization (<6 months vs 6 months to 2 years). Common genetic single nucleotide polymorphisms for genes encoding proteins involved in pharmacokinetic and/or pharmacodynamic pathways for letrozole are analyzed in order to determine if these single nucleotide polymorphisms contribute to individual variation in toxicity and efficacy of letrozole therapy.

Quality of life is assessed as during the first randomization.

Patients are followed annually.

PROJECTED ACCRUAL: A total of 4,700 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed primary invasive breast carcinoma resected at time of original diagnosis

  * No ductal carcinoma in situ
* Axillary lymph node negative, positive, or unknown
* No evidence of metastases
* No localized or distant breast cancer recurrence
* Not registered on protocol NCCTG-893052, any other IBCSG protocol, or protocol SWOG-S9623
* Hormone receptor status:

  * Estrogen or progesterone receptor positive as defined by tumor receptor content at least 10 fmol/mg protein or receptor positive by ERICA or PgRICA
  * Unknown status allowed if effort to determine status has been made by immunocytochemistry
* No contralateral breast cancer

PATIENT CHARACTERISTICS:

Age:

* Postmenopausal

Sex:

* Female

Menopausal status:

* Postmenopausal defined by one of the following:

  * Age 50 or over at start of adjuvant tamoxifen
  * Under age 50 and considered postmenopausal by treating physician at start of adjuvant tamoxifen
  * Under age 50 at start of adjuvant tamoxifen and had bilateral oophorectomy (surgical or radiation)
  * Under age 50 and premenopausal at start of adjuvant tamoxifen, but became amenorrheic during tamoxifen and remained amenorrheic for at least 1 year
  * Considered postmenopausal by physician with LH/FSH levels under the treatment center's postmenopausal limits

Performance status:

* ECOG 0-2

Life expectancy:

* At least 5 years

Hematopoietic:

* WBC ≥ 3,000/mm^3 OR
* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic:

* AST and/or ALT < 2 times upper limit of normal (ULN) (unless imaging examinations have ruled out metastatic disease)
* Alkaline phosphatase < 2 times ULN (unless imaging examinations have ruled out metastatic disease)

Renal:

* Not specified

Other:

* No concurrent medical or psychiatric condition that would preclude study participation
* No other malignancy within the past 5 years except adequately treated superficial squamous cell or basal cell skin cancer or carcinoma in situ of the cervix
* Able to swallow study drug
* Adequate oral intake

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior adjuvant chemotherapy allowed
* No concurrent chemotherapy

Endocrine therapy:

* Completed at least 4.5 but no more than 6 years of adjuvant tamoxifen after resection
* Completed at least 4.5-6 years of adjuvant aromatase inhibitor as initial therapy or after tamoxifen
* No more than 3 months since prior adjuvant tamoxifen
* No concurrent hormone replacement therapy (e.g., megestrol)
* No concurrent selective estrogen-receptor modulators (e.g., raloxifene or idoxifene)
* Concurrent intermittent vaginal estrogens (e.g., Estring) allowed if other local measures for intractable vaginal atrophy are insufficient
* No other concurrent aromatase inhibitors
* No more than 2 years since prior aromatase inhibitor therapy (re-randomization)

Radiotherapy:

* Prior radiotherapy allowed

Surgery:

* See Disease Characteristics

Other:

* At least 1 month since prior investigational drugs
* Prior treatment on a clinical trial for breast cancer allowed if permission has been obtained from the sponsors of the original study for their patient to participate on MA.17/JMA.17/BIG-97-01
* No prior placebo on core protocol
* No concurrent anticancer therapy
* Concurrent thyroid medication, calcium, vitamin D, and bisphosphonates allowed

Ages: 0 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5187 (Actual)
Dates: Start 1998-08-24 (Actual); Primary Completion 2003-08-22 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul E. Goss, MD, PhD, Study Chair — Massachusetts General Hospital; James N. Ingle, MD, Study Chair — Mayo Clinic; Monica Castiglione-Gertsch, MD, Study Chair — Insel Gruppe AG, University Hospital Bern; Nicholas J. Robert, MD, Study Chair — Fairfax Northern Virginia Hematology Oncology, PC - Fairfax; Silvana Martino, DO, Study Chair — Saint John's Cancer Institute; Hyman B. Muss, MD, Study Chair — University of Vermont; Martine J. Piccart-Gebhart, MD, PhD, Study Chair — Jules Bordet Institute
Locations (57):
- Canada (53):
  - Lethbridge Cancer Centre, Lethbridge, Alberta
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - NRGH - Nanaimo Cancer Clinic, Nanaimo, British Columbia
  - Penticton Regional Hospital, Penticton, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - BCCA - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - The Vitalite Health Network - Dr. Leon Richard, Moncton, New Brunswick
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - The Royal Victoria Hospital, Barrie, Ontario
  - Regional Cancer Program of the Hopital Regional, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Peterborough Regional Health Centre, Peterborough, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - North York General Hospital, Toronto, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Univ. Health Network-The Toronto General Hospital, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario
  - Trillium Health Centre - West Toronto, Toronto, Ontario
  - Humber River Regional Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - PEI Cancer Treatment Centre,Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - Centre de Sante et de services sociaux de Gatineau, Gatineau, Quebec
  - L'Hotel-Dieu de Levis, Lévis, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - CHUM - Hotel Dieu du Montreal, Montreal, Quebec
  - CHUM - Pavillon Saint-Luc, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec
  - CHA-Hopital Du St-Sacrement, Québec, Quebec
  - University Institute of Cardiology and, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- United Kingdom (4):
  - The Royal Marsden NHS Foundation Trust, London
  - Wythenshawe Hospital, Manchester
  - Christie's Hospital NHS Trust, Manchester
  - The Royal Marsden NHS Foundation Trust - Sutton, Surrey

REFERENCES:
- [Background] Baum M. Adjuvant endocrine therapy in postmenopausal women with early breast cancer: where are we now? Eur J Cancer. 2005 Aug;41(12):1667-77. doi: 10.1016/j.ejca.2005.05.006. PMID 16046117
- [Background] Baum M. Current status of aromatase inhibitors in the management of breast cancer and critique of the NCIC MA-17 trial. Cancer Control. 2004 Jul-Aug;11(4):217-21. doi: 10.1177/107327480401100402. PMID 15284712
- [Background] Booth CM, Pater JL, Goss PE. Identifying breast cancer patients most likely to benefit from aromatase inhibitor therapy after adjuvant tamoxifen. Cancer. 2007 May 1;109(9):1927-8; author reply 1928. doi: 10.1002/cncr.22613. No abstract available. PMID 17354227
- [Background] Buzdar A, Chlebowski R, Cuzick J, Duffy S, Forbes J, Jonat W, Ravdin P. Defining the role of aromatase inhibitors in the adjuvant endocrine treatment of early breast cancer. Curr Med Res Opin. 2006 Aug;22(8):1575-85. doi: 10.1185/030079906X120940. PMID 16870082
- [Background] Scott LJ, Keam SJ. Letrozole : in postmenopausal hormone-responsive early-stage breast cancer. Drugs. 2006;66(3):353-62. doi: 10.2165/00003495-200666030-00010. PMID 16526826
- [Background] Vakaet L. Re: Randomized trial of letrozole following tamoxifen as extended adjuvant therapy in receptor-positive breast cancer: updated findings from NCIC CTG MA.17. J Natl Cancer Inst. 2006 Aug 16;98(16):1162; author reply 1162-3. doi: 10.1093/jnci/djj323. No abstract available. PMID 16912269
- [Background] Wardley AM. Emerging data on optimal adjuvant endocrine therapy: Breast International Group trial 1-98/MA.17. Clin Breast Cancer. 2006 Feb;6 Suppl 2:S45-50. doi: 10.3816/cbc.2006.s.003. PMID 16595026
- [Result] Goss PE, Ingle JN, Martino S, et al.: Outcomes of women who were premenopausal at diagnosis of early stage breast cancer in the NCIC CTG MA17 trial. [Abstract] 32nd Annual San Antonio Breast Cancer Symposium, December 9-13, 2009, San Antonio, Texas. A-13, 2009.
- [Result] Goss PE, Ingle JN, Pater JL, Martino S, Robert NJ, Muss HB, Piccart MJ, Castiglione M, Shepherd LE, Pritchard KI, Livingston RB, Davidson NE, Norton L, Perez EA, Abrams JS, Cameron DA, Palmer MJ, Tu D. Late extended adjuvant treatment with letrozole improves outcome in women with early-stage breast cancer who complete 5 years of tamoxifen. J Clin Oncol. 2008 Apr 20;26(12):1948-55. doi: 10.1200/JCO.2007.11.6798. Epub 2008 Mar 10. PMID 18332475
- [Result] Ingle JN, Tu D, Pater JL, Muss HB, Martino S, Robert NJ, Piccart MJ, Castiglione M, Shepherd LE, Pritchard KI, Livingston RB, Davidson NE, Norton L, Perez EA, Abrams JS, Cameron DA, Palmer MJ, Goss PE. Intent-to-treat analysis of the placebo-controlled trial of letrozole for extended adjuvant therapy in early breast cancer: NCIC CTG MA.17. Ann Oncol. 2008 May;19(5):877-82. doi: 10.1093/annonc/mdm566. Epub 2008 Mar 10. PMID 18332043
- [Result] Muss HB, Tu D, Ingle JN, Martino S, Robert NJ, Pater JL, Whelan TJ, Palmer MJ, Piccart MJ, Shepherd LE, Pritchard KI, He Z, Goss PE. Efficacy, toxicity, and quality of life in older women with early-stage breast cancer treated with letrozole or placebo after 5 years of tamoxifen: NCIC CTG intergroup trial MA.17. J Clin Oncol. 2008 Apr 20;26(12):1956-64. doi: 10.1200/JCO.2007.12.6334. Epub 2008 Mar 10. PMID 18332474
- [Result] Chapman JW, Meng D, Shepherd L, et al.: Competing causes of death in breast cancer extended adjuvant endocrine therapy: NCIC CTG MA.17. [Abstract] American Society of Clinical Oncology 2007 Breast Cancer Symposium, 7-8 September 2007, San Francisco, California A-56, 2007.
- [Result] Goss PE, Ingle JN, Martino S, Robert NJ, Muss HB, Piccart MJ, Castiglione M, Tu D, Shepherd LE, Pritchard KI, Livingston RB, Davidson NE, Norton L, Perez EA, Abrams JS, Cameron DA, Palmer MJ, Pater JL; National Cancer Institute of Canada Clinical Trials Group MA.17. Efficacy of letrozole extended adjuvant therapy according to estrogen receptor and progesterone receptor status of the primary tumor: National Cancer Institute of Canada Clinical Trials Group MA.17. J Clin Oncol. 2007 May 20;25(15):2006-11. doi: 10.1200/JCO.2006.09.4482. Epub 2007 Apr 23. PMID 17452676
- [Result] Goss P: Breaking the 5-year barrier: results from the MA.17 extended adjuvant trial in women who have completed adjuvant tamoxifen treatment. [Abstract] European Journal of Cancer Supplements 4 (9): 10-5, 2006.
- [Result] Ingle JN, Tu D, Pater JL, Martino S, Robert NJ, Muss HB, Piccart MJ, Castiglione M, Shepherd LE, Pritchard KI, Livingston RB, Davidson NE, Norton L, Perez EA, Abrams JS, Cameron DA, Palmer MJ, Goss PE. Duration of letrozole treatment and outcomes in the placebo-controlled NCIC CTG MA.17 extended adjuvant therapy trial. Breast Cancer Res Treat. 2006 Oct;99(3):295-300. doi: 10.1007/s10549-006-9207-y. Epub 2006 Mar 16. PMID 16541302
- [Result] Ingle J, Tu D, Shepherd L, et al.: NCIC CTG MA.17: intent to treat analysis (ITT) of randomized patients after a median follow-up of 54 months. [Abstract] J Clin Oncol 24 (Suppl 18): A-549, 2006.
- [Result] Moy B, Tu D, Shepherd LE, et al.: NCIC CTG MA.17: tolerability of letrozole among ethnic minority women. [Abstract] J Clin Oncol 24 (Suppl 18): A-6018, 305s, 2006.
- [Result] Pater JL, Tu D, Ingle JN, et al.: An evaluation of the early termination (ET) of MA.17 extended adjuvant therapy trial. [Abstract] Breast Cancer Res Treat 100 (Suppl 1): A-2081, S107-8, 2006.
- [Result] Perez EA, Josse RG, Pritchard KI, Ingle JN, Martino S, Findlay BP, Shenkier TN, Tozer RG, Palmer MJ, Shepherd LE, Liu S, Tu D, Goss PE. Effect of letrozole versus placebo on bone mineral density in women with primary breast cancer completing 5 or more years of adjuvant tamoxifen: a companion study to NCIC CTG MA.17. J Clin Oncol. 2006 Aug 1;24(22):3629-35. doi: 10.1200/JCO.2005.05.4882. Epub 2006 Jul 5. PMID 16822845
- [Result] Robert NJ, Goss PE, Ingle JN, et al.: Updated analysis of NCIC CTG MA.17 (letrozole vs. placebo to letrozole vs placebo) post unblinding. [Abstract] J Clin Oncol 24 (Suppl 18): A-550, 2006.
- [Result] Abetz L, Barghout V, Thomas S, et al.: Letrozole did not worsen quality of life relative to placebo in post-menopausal women with early breast cancer: results from the US subjects of the MA-17 study. [Abstract] Breast Cancer Research and Treatment 94 (Suppl 1): A-2047, 2005.
- [Result] Goss PE, Ingle JN, Martino S, Robert NJ, Muss HB, Piccart MJ, Castiglione M, Tu D, Shepherd LE, Pritchard KI, Livingston RB, Davidson NE, Norton L, Perez EA, Abrams JS, Cameron DA, Palmer MJ, Pater JL. Randomized trial of letrozole following tamoxifen as extended adjuvant therapy in receptor-positive breast cancer: updated findings from NCIC CTG MA.17. J Natl Cancer Inst. 2005 Sep 7;97(17):1262-71. doi: 10.1093/jnci/dji250. PMID 16145047
- [Result] Goss PE, Ingle JN, Palmer MJ, et al.: Updated analysis of NCIC CTG MA.17 (letrozole vs. placebo to letrozole vs placebo) post unblinding. [Abstract] Breast Cancer Research and Treatment 94 (Suppl 1): A-16, 2005.
- [Result] Goss PE, Ingle JN, Tu D: NCIC CTG MA17: disease free survival according to estrogen receptor and progesterone receptor status of the primary tumor. [Abstract] Breast Cancer Research and Treatment 94 (Suppl 1): A-2042, 2005.
- [Result] Ingle JN, Goss PE, Tu D: Analysis of duration of letrozole extended adjuvant therapy as measured by hazard ratios of disease recurrence over time for patients on NCIC CTG MA.17. [Abstract] Breast Cancer Research and Treatment 94 (Suppl 1): A-17, 2005.
- [Result] Luk C, Goss P, Pritchard K, et al.: Determinants of preferences for starting extended adjuvant letrozole (L) in postmenopausal women following five years of tamoxifen. [Abstract] J Clin Oncol 23 (Suppl 16): A-642, 39s, 2005.
- [Result] Vachon CM, Ingle JN, Scott CG, et al.: Pilot study of changes in mammographic density in women treated with letrozole or placebo on NCIC CTG MA17. [Abstract] Breast Cancer Research and Treatment 94 (Suppl 1): A-6005, 2005.
- [Result] Whelan TJ, Goss PE, Ingle JN, Pater JL, Tu D, Pritchard K, Liu S, Shepherd LE, Palmer M, Robert NJ, Martino S, Muss HB. Assessment of quality of life in MA.17: a randomized, placebo-controlled trial of letrozole after 5 years of tamoxifen in postmenopausal women. J Clin Oncol. 2005 Oct 1;23(28):6931-40. doi: 10.1200/JCO.2005.11.181. Epub 2005 Sep 12. PMID 16157934
- [Result] Goss PE, Ingle JN, Martino S, et al.: Updated analysis of the NCIC CTG MA.17 randomized placebo (P) controlled trial of letrozole (L) after five years of tamoxifen in postmenopausal women with early stage breast cancer. [Abstract] J Clin Oncol 22 (Suppl 14): A-847, 88s, 2004.
- [Result] Goss PE, Ingle JN, Martino S, Robert NJ, Muss HB, Piccart MJ, Castiglione M, Tu D, Shepherd LE, Pritchard KI, Livingston RB, Davidson NE, Norton L, Perez EA, Abrams JS, Therasse P, Palmer MJ, Pater JL. A randomized trial of letrozole in postmenopausal women after five years of tamoxifen therapy for early-stage breast cancer. N Engl J Med. 2003 Nov 6;349(19):1793-802. doi: 10.1056/NEJMoa032312. Epub 2003 Oct 9. PMID 14551341
- [Derived] Ethier JL, Anderson GM, Austin PC, Clemons M, Parulekar W, Shepherd L, Summers Trasiewicz L, Tu D, Amir E. Influence of the competing risk of death on estimates of disease recurrence in trials of adjuvant endocrine therapy for early-stage breast cancer: A secondary analysis of MA.27, MA.17 and MA.17R. Eur J Cancer. 2021 May;149:117-127. doi: 10.1016/j.ejca.2021.02.034. Epub 2021 Apr 11. PMID 33853037
- [Derived] Goss PE, Ingle JN, Pritchard KI, Robert NJ, Muss H, Gralow J, Gelmon K, Whelan T, Strasser-Weippl K, Rubin S, Sturtz K, Wolff AC, Winer E, Hudis C, Stopeck A, Beck JT, Kaur JS, Whelan K, Tu D, Parulekar WR. Extending Aromatase-Inhibitor Adjuvant Therapy to 10 Years. N Engl J Med. 2016 Jul 21;375(3):209-19. doi: 10.1056/NEJMoa1604700. Epub 2016 Jun 5. PMID 27264120